CLINICAL TRIAL: NCT00512057
Title: APEX Study: Effects of Allopurinol on Coronary and Peripheral Endothelial Function in Patients With Cardiac Syndrome X
Acronym: APEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Chim Lang, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: apex001 version6
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-02

CONDITIONS: Syndrome X
Keywords: cardiac syndrome X; endothelial function
MeSH Terms: conditions — Microvascular Angina | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: allopurinol
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: allopurinol — allopurinol 300mg twice a day
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Morbidity of patients with cardiac syndrome X (typical anginal-like chest pain and normal coronary arteriograms) is high with continuing episodes of chest pain and frequent hospital readmissions. Management of this syndrome represents a major challenge to the treating physician. Evidence for the important role of endothelial dysfunction and oxidative stress in the pathogenesis of cardiac syndrome X has been recently strengthened by the finding that basal superoxide production predicts future cardiovascular events in this patient group. The investigators have recently shown that high-dose allopurinol abolishes vascular oxidative stress and improves endothelial function in patients with chronic heart failure, which makes allopurinol a prime candidate to reduce oxidative stress in syndrome X. The hypothesis to be tested in this study is whether allopurinol offers dual benefits of improving vascular function and reducing myocardial ischaemia in patients with cardiac syndrome X. This study may discover a novel way to improve endothelial function and anginal symptoms which are often debilitating in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Typical history of angina
* Positive exercise treadmill test and normal coronary angiogram

Exclusion Criteria:

* Significant valvular heart disease or left ventricular hypertrophy
* Age <18 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate the effects of allopurinol on coronary and peripheral microvascular and endothelial function in patients with cardiac syndrome X | 3-5 years

SECONDARY OUTCOMES:
The secondary objectives of this study are to assess the effects of allopurinol on chest pain incidence, maximal ST-segment depression and Duke's score | 3- 5years

CONTACTS AND LOCATIONS:
Overall Officials: Chim Lang, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Dundee, United Kingdom